CLINICAL TRIAL: NCT01150903
Title: Prevalence and Incidence of Underlying Disease Diagnosed in Men With Erectile Dysfunction When Prescribed a PDE5i for the First Time
Brief Title: Identification of Underlying Conditions in Men Prescribed a PDE5 Inhibitor
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A1481287
Record Dates: First submitted 2010-06-24; First posted 2010-06-25 (Estimated); Results first posted 2012-05-11 (Estimated); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Erectile Dysfunction; Cardiovascular Diseases; Male Urogenital Diseases
Keywords: erectile dysfunction; phosphodiesterase inhibitor; cardiovascular diseases
MeSH Terms: conditions — Erectile Dysfunction; Cardiovascular Diseases; Male Urogenital Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PDE5 inhibitor prescription
  Interventions: Other: no intervention
- Age-matched Control
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — non-interventional study
  Groups: PDE5 inhibitor prescription
Other: no intervention — non-interventional study
  Groups: Age-matched Control

SUMMARY:
Erectile dysfunction (ED) has been identified as an independent risk factor for existing cardiovascular disease, preceding a major cardiovascular event by an average of about 5 years. Are men prescribed a PDE5 inhibitor for ED more likely to have a new diagnosis of underlying medical conditions compared to men of a similar age not receiving PDE5 inhibitor treatment?

ELIGIBILITY:
Inclusion Criteria:

* Records of men aged >18 years with an index PDE5 inhibitor (sildenafil, tadalafil or vardenafil) prescription between January 1st, 1999, and June 30th, 2008
* no prior PDE5 inhibitor prescription before the index prescription
* continuous enrolment with medical history for ≥60 months prior to the index prescription date

Exclusion Criteria:

* Records of female subjects and any male subjects not meeting the inclusion criteria will be excluded
* A subject can only be selected once independent of the assignment to the target or the control populations.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a PDE5 inhibitor prescription and within the age-match control.
Sampling Method: Non-Probability Sample
Enrollment: 98832 (Actual)
Dates: Start 2010-05; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- [Derived] Kirby MG, Schnetzler G, Zou KH, Symonds T. Prevalence and detection rate of underlying disease in men with erectile dysfunction receiving phosphodiesterase type 5 inhibitors in the United Kingdom: a retrospective database study. Int J Clin Pract. 2011 Jul;65(7):797-806. doi: 10.1111/j.1742-1241.2011.02693.x. PMID 21676121
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481287&StudyName=Identification%20of%20underlying%20conditions%20in%20men%20prescribed%20a%20PDE5%20inhibitor%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Index PDE5i Prescription: Participants who received index phosphodiesterase type 5 inhibitor (PDE5i) (sildenafil, tadalafil or vardenafil) prescription between January 1, 1999 and June 30, 2008, as identified from the United Kingdom - The Health Improvement Network (UK-THIN) database (target population).
- Control (Without PDE5i Prescription): Age-matched participants without any PDE5i (sildenafil, tadalafil or vardenafil) prescription between January 1, 1999 and June 30, 2008, as identified from the UK-THIN database (control population).
Period: Overall Study
Arm/Group | Index PDE5i Prescription | Control (Without PDE5i Prescription)
Started | 24708 | 74124
Completed | 24708 | 74124
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Index PDE5i Prescription | Control (Without PDE5i Prescription) | Total
Number analyzed (Participants) | 24708 | 74124 | 98832
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.63 (11.59) | 57.63 (11.59) | 57.63 (11.59)
Age, Continuous [Median (Full Range); unit: Years] | 59.0 [18.0 to 91.0] | 59.0 [18.0 to 91.0] | 59.0 [18.0 to 91.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 24708 | 74124 | 98832

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Underlying Condition Until Day -1 of the Index PDE5i Prescription
Description: Underlying conditions were defined as any diagnosis of interest recorded in the relevant time period. Diagnoses of interest were coded and categorized in to vasculogenic, urologic, neurogenic, hormonal, drug induced and psychogenic disorders.
Time Frame: Day -92 up to Day -1 of index prescription
Population: Evaluable analysis population included all participants who received an index PDE5i prescription (sildenafil, tadalafil or vardenafil) during the study period (target population) and age-matched participants without any PDE5i prescription during the study period (control population). Last observation carried forward method was used.
Measure: Number; unit: Percentage of participants
Arm/Group | Index PDE5i Prescription | Control (Without PDE5i Prescription)
Number analyzed (Participants) | 24708 | 74124
Percentage of participants | 70.23 | 55.73
Statistical Analysis 1: Comparison: Index PDE5i Prescription vs Control (Without PDE5i Prescription); Chi-square test was used to calculate p-value; Test type: Superiority or Other; p < 0.001, Chi-squared

2. Primary Outcome: Cumulative Percentage of Participants With New Diagnosis of Underlying Condition Between Index PDE5i Prescription (Day 0) and Day 91
Description: New diagnosis of underlying condition at prescription was defined as any new diagnosis of interest recorded in the relevant time period. Diagnoses of interest were coded and categorized in to vasculogenic, urologic, neurogenic, hormonal, drug induced and psychogenic disorders.
Time Frame: Day 0 to Day 91 post index prescription
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Index PDE5i Prescription | Control (Without PDE5i Prescription)
Number analyzed (Participants) | 24708 | 74124
Percentage of participants | 11.53 | 7.49
Statistical Analysis 1: Comparison: Index PDE5i Prescription vs Control (Without PDE5i Prescription); Chi-square test was used to calculate p-value; Test type: Superiority or Other; p < 0.001, Chi-squared

3. Primary Outcome: Percentage of Participants With New Diagnosis of Underlying Condition Between Day -92 and Day -1 Prior to the Index PDE5i Prescription
Description: New diagnosis of underlying condition was defined as any new diagnosis of interest recorded in the relevant time period. Diagnoses of interest were coded and categorized in to vasculogenic, urologic, neurogenic, hormonal, drug induced and psychogenic disorders.
Time Frame: Day -92 up to Day -1 of index prescription
Population: Evaluable analysis population included all participants who received an index PDE5i prescription (sildenafil, tadalafil or vardenafil) during the study period (target population). Last observation carried forward method was used.
Measure: Number; unit: Percentage of participants
Arm/Group | Index PDE5i Prescription
Number analyzed (Participants) | 24708
Percentage of participants | 11.08

4. Primary Outcome: Percentage of Participants With New Diagnosis of Underlying Condition Between Day 366 and Day 457 Post the Index PDE5i Prescription
Description: as for outcome 3
Time Frame: Day 366 up to Day 457 post index prescription
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Index PDE5i Prescription
Number analyzed (Participants) | 24708
Percentage of participants | 5.65

5. Primary Outcome: Percentage of Participants With Underlying Condition at PDE5i Market Introduction During the Early Study Period
Description: Underlying condition at PDE5i market introduction was defined as any diagnosis of interest until day -1 in participants who received the index prescription between January 1, 1999 and December 31, 2001 for the three years period combined. Diagnoses of interest were coded and categorized in to vasculogenic, urologic, neurogenic, hormonal, drug induced and psychogenic disorders.
Time Frame: Up to 3 years (Early study period - January 1999 to December 2001)
Population: Evaluable analysis population included all participants who received an index PDE5i prescription (sildenafil, tadalafil or vardenafil) during the study period (target population). Last observation carried forward method was used. Here, the 'N' (number of participants analyzed) is signifying those participants who were evaluable for this measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Index PDE5i Prescription
Number analyzed (Participants) | 892
Percentage of participants | 67.49

6. Secondary Outcome: Percentage of Participants With New Diagnosis of Underlying Condition at PDE5i Market Introduction During the Early Study Period
Description: New diagnosis of underlying condition at PDE5i market introduction was defined as any new diagnosis of interest until day -1 in participants who received the index prescription between January 1, 1999 and December 31, 2001 for the three years period combined. Diagnoses of interest were coded and categorized in to vasculogenic, urologic, neurogenic, hormonal, drug induced and psychogenic disorders.
Time Frame: Up to 3 years (Early study period - January 1999 to December 2001)
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Index PDE5i Prescription
Number analyzed (Participants) | 892
Percentage of participants | 11.32

7. Secondary Outcome: Percentage of Participants With Underlying Condition at PDE5i Establishment During the End of Study Period
Description: Underlying condition at PDE5i market introduction was defined as any diagnosis of interest until day -1 in participants who received the index prescription between July 1, 2006 and June 30, 2008 for the two years period combined. Diagnoses of interest were coded and categorized in to vasculogenic, urologic, neurogenic, hormonal, drug induced and psychogenic disorders.
Time Frame: Up to 2 years (End of study period - July 2006 to June 2008)
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Index PDE5i Prescription
Number analyzed (Participants) | 9862
Percentage of participants | 72.14

8. Secondary Outcome: Percentage of Participants With New Diagnosis of Underlying Condition at PDE5i Establishment During the End of Study Period
Description: New diagnosis of underlying condition at PDE5i establishment was defined as any new diagnosis of interest between day 0 (index prescription) and day 91 in participants who received the index prescription between July 1, 2006 and June 30, 2008 for the two-years period combined. Diagnoses of interest were coded and categorized in to vasculogenic, urologic, neurogenic, hormonal, drug induced and psychogenic disorders.
Time Frame: Up to 2 years (End of study period - July 2006 to June 2008)
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Index PDE5i Prescription
Number analyzed (Participants) | 9862
Percentage of participants | 11.06

ADVERSE EVENTS:
Description: As it was a retrospective study and no safety data (adverse events and serious adverse events) were analyzed, hence number of participants affected and at risk were reported as 0.
Arm/Group | Index PDE5i Prescription | Control (Without PDE5i Prescription)
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.